CLINICAL TRIAL: NCT05932108
Title: Evaluation of the Violence Prevention Initiative TERMA in Forensic Psychiatric Inpatient Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: TERMA
Record Dates: First submitted 2023-06-15; First posted 2023-07-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Forensic Nursing; Forensic Psychiatry
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Staff: Educational intervention in TERMA. All staff are required to attend the education.
  Interventions: Behavioral: Education in TERMA
- Patients: Patients will not attend any education in TERMA. Data will be collected before and after the staffs education to se if the patients think the attitude of the staff have changed.
  Interventions: Other: Changed work routines based on TERMA

INTERVENTIONS:
Behavioral: Education in TERMA — Education of staff in TERMA. The primary aim of TERMA is to prevent aggression and violence through a system of low-effective treatment that is divided into escalating levels based on the patient's aggression level, risk of violence, and acts of violence . The TERMA model focuses on treatment, communication, and management of compassionate healthcare in forensic psychiatric settings . The levels of the TERMA model are in a "cascading" order, whereby if the treatment and management of one level are ineffective, the next level is initiated, and so on. The primary level involves the daily behavior and health status of the patient. The secondary level involves risk assessment and violence management, with a focus on creating an understanding of the situation for both the patient and healthcare workers. The tertiary level is utilized when violence cannot be avoided . Each level corresponds to a specific response according to the demands of the situation and environment.
  Groups: Staff
Other: Changed work routines based on TERMA — NO planned intervention but staff work routines and behavior may change after their education in TERMA. Patients are exposed to these changes.
  Groups: Patients

SUMMARY:
The aim of this project is to evaluate the violence prevention method Therapeutic meeting with aggression (TERMA) regarding adverse events and perceived safety by patients and staff within forensic psychiatric inpatient care. Additionally, the project will investigate whether the organizational culture influences the implementation of the TERMA method and the experiences of patients and staff in situations involving threats, violence, and the use of coercive measures.

DETAILED DESCRIPTION:
Overall aim The aim of this project is to evaluate the violence prevention method Therapeutic meeting with aggression (TERMA) regarding adverse events and perceived safety by patients and staff within forensic psychiatric inpatient care. Additionally, the project will investigate whether the organizational culture influences the implementation of the TERMA method and the experiences of patients and staff in situations involving threats, violence, and the use of coercive measures.

Research questions

* To what extent does the implementation of TERMA impact the perceived safety of staff and patients in a forensic psychiatric inpatient setting, as measured by the Perceived Safety Questionnaire (E13)?
* What is the effect of implementing TERMA on the frequency of incidents of aggression and violence, healthcare and occupational injuries, and the use of coercive measures in a forensic psychiatric inpatient setting?
* How does the implementation of TERMA impact the organizational culture of a forensic psychiatric inpatient unit, as measured by changes in perceived safety, incidents of aggression and violence, healthcare and occupational injuries, and the use of coercive measures, as assessed by the Organisations Value Questionnaire (OVQ) questionnaire?
* How do patients perceive threatening and violent situations, exposure to coercive measures, and the implementation of TERMA in a forensic psychiatric inpatient setting?
* What are the attitudes and perceptions of staff towards working with TERMA, how do they respond to threatening and violent situations, and what is the impact of these factors on the work environment in a forensic psychiatric inpatient setting? Introduction Forensic psychiatric care is provided to patients who have been convicted of a crime that was perpetrated while having a severe mental disorder. Severe mental illness is a judicial concept within Swedish law and is not a medical diagnosis. The primary goal of forensic psychiatric care is to rehabilitate the patients so they can be reintegrated into society without risk of committing new crimes. Swedish law states that health care should strive to protect and strengthen the integrity and participation of the patient. This is, however, difficult within forensic psychiatric care, which is not voluntarily, involves mandatory treatment and deprives patients of liberty. Maintaining a therapeutic relationship with patients, while managing their reactions and emotions in high-security wards, can be challenging.

Forensic psychiatric patients are a heterogeneous group, given their various psycho pathologies, criminal histories and risk factors for reoffending. Patients sentenced to forensic psychiatric care are under involuntary care for long periods of time and rehabilitation length of 5-6 years are not unusual. Aggressive and violent behavior among patients is a prevalent occurrence in forensic psychiatry and a hindrance for successful rehabilitation. The complex composition of mental illnesses contributes to an experience of an insecure environment for both patients and healthcare personnel.

There is a need for research on the content and effects of managing aggression and violence. Several methods have been developed to manage and prevent such behaviors. One such method is the Therapeutic Meeting with Aggression (TERMA). It has previously been implemented in inpatient forensic psychiatric care in Sweden but further research is needed in evaluating its usefulness.

Therapeutic meeting with aggression (TERMA) TERMA was developed from the Norwegian Bergen model, with modifications made to align with the Swedish healthcare and legal systems. The primary aim of TERMA is to prevent aggression and violence through a system of low-effective treatment that is divided into escalating levels based on the patient's aggression level, risk of violence, and acts of violence. The TERMA model focuses on treatment, communication, and management of compassionate healthcare in forensic psychiatric settings. The levels of the TERMA model are in a "cascading" order, whereby if the treatment and management of one level are ineffective, the next level is initiated, and so on. The primary level involves the daily behavior and health status of the patient. The secondary level involves risk assessment and violence management, with a focus on creating an understanding of the situation for both the patient and healthcare workers. The tertiary level is utilized when violence cannot be avoided. Each level corresponds to a specific response according to the demands of the situation and environment.

ELIGIBILITY:
Inclusion Criteria Staff:

* ≥ 18 years of age who
* work in forensic psychiatric inpatient care,
* understand and speak Swedish or English, and are
* willing to participate and sign a consent form.

Exclusion Criteria Staff:

* not willing to participate

Inclusion Criteria Patients:

* ≥ 18 years of age who are
* admitted to forensic psychiatric inpatient care according to the Swedish Forensic Psychiatric Care Act,
* understand and speak Swedish or English,
* have approval to participate from the treating physician, and are
* willing to participate and sign a consent form.

Exclusion Criteria Patients:

* not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Staff at a forensic psychiatry department. Patients at a forensic psychiatry departmen
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Perceived Safety Questionnaire (E13) | Change measure (baseline to 6 months)
  Questionnaire data on perceived safety. E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.
Perceived Safety Questionnaire (E13) | Change measure (baseline to 1 year)
  Questionnaire data on perceived safety. E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.

SECONDARY OUTCOMES:
Organisations Value Questionnaire (OVQ). | Change measure (baseline to 6 months)
  Questionnaire data on organizational culture. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
Organisations Value Questionnaire (OVQ). | Change measure (baseline to 1 year)
  Questionnaire data on organizational culture. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
Organisations Value Questionnaire (OVQ)_Safety Questionnaire (E13) | Baseline
  Correlation between organizational culture and perceived safety. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
  E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.
Organisations Value Questionnaire (OVQ)_Safety Questionnaire (E13) | 6 months
  Correlation between organizational culture and perceived safety. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
  E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.
Organisations Value Questionnaire (OVQ)_Safety Questionnaire (E13) | 1 year
  Correlation between organizational culture and perceived safety. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
  E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.
Organisations Value Questionnaire (OVQ)_Safety Questionnaire (E13) | Baseline (OVQ) and 6 months (E13)
  Correlation between organizational culture and perceived safety. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
  E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.
Organisations Value Questionnaire (OVQ)_Safety Questionnaire (E13) | Baseline (OVQ) and 1 year (E13)
  Correlation between organizational culture and perceived safety. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
  E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.
Organisations Value Questionnaire (OVQ)_Safety Questionnaire (E13) | Baseline (OVQ) and change in E13 (baseline to 6 months)
  Correlation between organizational culture and perceived safety. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
  E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.
Organisations Value Questionnaire (OVQ)_Safety Questionnaire (E13) | Baseline (OVQ) and change in E13 (baseline to 1 year)
  Correlation between organizational culture and perceived safety. OVQ is used to measure the the overall organizational culture and dimensions human relation (HR), open systems (OS), rational goal (RG) and internal process (IP). It consisted of 52 items with alternative answers of the Likert type ranging from "strongly disagree" to "strongly agree". Averages were calculated for the total OVQ and for each subscale; a high score indicates strong disagreement. Minimum value 52, maximum value 520 for the total OVQ. Minimum value 13, maximum value 130 for each of the subscales.
  E13 measures factors such as self-estimated safety, feeling of safety, acts of violence and coercion, reaction and aggression measurements and cause of aggression in the wards. The questionnaire consists of 13 statements whose agreement is answered on a four-point Likert scale from completely agree to completely disagree. Minimum value=13, maximum value=52, higher values means better outcome.
Number of coercive measures | From 1 year before baseline to 1 year after study end
  Data from medical records on coercive measures, for example restraint and forced medication
Incidence of threat and violence | From 1 year before baseline to 1 year after study end
  Deviation reports from the incidence report system "MedControl PRO"

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wallström, PhD, Principal Investigator — Västra Götalandsregionen

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD)